CLINICAL TRIAL: NCT04717544
Title: Embedding Comprehensive Smoking Cessation Programs Into Community Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: University of California (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 28CP-0040
Record Dates: First submitted 2021-01-04; First posted 2021-01-22 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Implementation; Sustainable
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Active Comparator): Healthcare providers from clinics participating in the intervention refer existing clients to study coordinators for smoking cessation services, wherein the coordinators link clients to the smoking cessation services, which include: 1) a weekly cognitive-behavioral therapy smoking cessation (CBT) counseling group; and 2) smoking cessation medication, which include varenicline (Chantix), bupropion (Zyban) and nicotine patches, gum, and lozenges. Clients interested in these medications will meet with the prescribing clinician to help choose the best prescription option.
  In addition to linking clients to the smoking cessation services, coordinators will invite clients to participate in the outcome study.
  Existing clients can sign-up for these services and/or the outcome study directly with the study coordinators and do not require a healthcare provider referral.
  Interventions: Behavioral: Intervention Arm
- Treatment As Usual Arm (No Intervention): Existing clients can be referred to the outcome study by their healthcare providers from clinics designated as TAU or they can sign-up directly with the study coordinators.

INTERVENTIONS:
Behavioral: Intervention Arm — The smoking cessation intervention will include 1) a six-week, 60-75 minute weekly cognitive-behavioral therapy (CBT) smoking cessation counseling group; and 2) smoking cessation medication include varenicline (Chantix), bupropion (Zyban) and nicotine replacement therapy (NRT). Dispensing these medications will include a 15-minute medication management visit with a prescribing clinician. Clients will choose their own preferred treatment. The standard prescription for NRT will include a transdermal patch at a dose that approximates for current average mg of nicotine intake and nicotine gums or lozenges (in either 2 mg or 4 mg strengths). Prescription for varenicline will be 0.5 mg once daily for three days, then 0.5 mg twice daily for the next four days, then 1 mg twice daily thereafter. Absent any contraindications to the drugs listed above, bupropion (Zyban) 150mg will be offered and prescribed once daily for one week, following by bupropion 300 mg once daily thereafter.
  Arms: Intervention Arm

SUMMARY:
The study will evaluate a sustainable tobacco screening, treatment intervention, and cessation program implemented within both Los Angeles County (LAC)-Department of Health Services (LACDHS)-operated outpatient primary care clinics and in LAC-Department of Mental Health (LACDMH)-operated community mental health clinics. This is a three year implementation study funded by the University of California Office of the President Tobacco Related Disease Research Program (TRDRP). This project will support the implementation of smoking cessation services delivered in LACDHS and LACDMH clinics and will evaluate the effectiveness and feasibility of these services.

DETAILED DESCRIPTION:
The research hypothesis is that training LACDHS and LACDMH staff and clinicians to screen for and treat tobacco use disorder will improve rates of remission from tobacco use disorder in the clients served by each system.

This is a cluster randomized comparative effectiveness trial that compares intervention clinics (offer smoking cessation group counseling and medication management) integrated into primary care and community mental health clinics with treatment as usual (offering information about the California Smoker's Helpline and informal provider counseling). The specific aim is to randomize 17 clinics (11 at LACDHS and 6 at LACDMH), with a 5:1 ratio in the assignment of clinical sites assigned to offer smoking cessation services as compared to the treatment as usual (TAU).

In addition to providing support for the implementation of the smoking cessation services, the study will enroll 1,200 clients with tobacco use disorder from all 17 participating clinics for an outcome study; 1000 people from clinical sites where smoking cessation treatment are being offered and 200 people with tobacco use disorder from the TAU clinical sites. The primary study outcome is to determine if there will be higher rates of smoking cessation in the implementation sites as compared with TAU sites that do not offer smoking cessation treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* smoke 3 or more cigarettes or cigars per day
* have thought about smoking cessation
* be enrolled in care at either LACDHS and/or LACDMH.

Exclusion Criteria:

* under 18 years
* smoke less than 3 cigarettes or cigars per day
* not interested in smoking cessation
* not enrolled in care at either LACDHS and/or LACDMH.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Smoking Cessation Rate | Change in carbon monoxide and cotinine levels from Baseline at 3 months
  The primary outcome is to determine if there will be higher rates of smoking cessation in the intervention sites as compared with matched non-intervention sites. In order to measure these rates, study participants will be asked to complete two objective measures collected at 3-month, 6-month and 12-month follow-up. These measures include a carbon monoxide breathalyzer (piCO+smokerlyzer) and urinary rapid dipstick cotinine test (NicCheck). A participant will count as having quit if they reported having abstained from smoking cigarettes/cigars for seven consecutive days and if this report is corroborated by carbon monoxide and cotinine testing.
Smoking Cessation Rate | Change in carbon monoxide and cotinine levels from 3 months at 6 months
  The primary outcome is to determine if there will be higher rates of smoking cessation in the intervention sites as compared with matched non-intervention sites. In order to measure these rates, study participants will be asked to complete two objective measures collected at 3-month, 6-month and 12-month follow-up. These measures include a carbon monoxide breathalyzer (piCO+smokerlyzer) and urinary rapid dipstick cotinine test (NicCheck). A participant will count as having quit if they reported having abstained from smoking cigarettes/cigars for seven consecutive days and if this report is corroborated by carbon monoxide and cotinine testing.
Smoking Cessation Rate | Change in carbon monoxide and cotinine levels from 6 months at 12 months
  The primary outcome is to determine if there will be higher rates of smoking cessation in the intervention sites as compared with matched non-intervention sites. In order to measure these rates, study participants will be asked to complete two objective measures collected at 3-month, 6-month and 12-month follow-up. These measures include a carbon monoxide breathalyzer (piCO+smokerlyzer) and urinary rapid dipstick cotinine test (NicCheck). A participant will count as having quit if they reported having abstained from smoking cigarettes/cigars for seven consecutive days and if this report is corroborated by carbon monoxide and cotinine testing.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore C Friedman, M.D., Ph.D., Principal Investigator — Charles R. Drew University of Medicine & Science
Locations (1):
- Los Angeles County Department of Health Services and Department of Mental Health Services, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meredith LR, Hurley B, Friedman TC, Lee ML, Rodriguez L, Lopez B, Mtume N, Dixon T, Belani HK, Hsieh S, Ray LA. Implementation of Specialty Tobacco Use Disorder Services in a Community Health Setting: Support for Enhanced Prescription Practices. J Addict Med. 2023 Nov-Dec 01;17(6):677-684. doi: 10.1097/ADM.0000000000001211. Epub 2023 Aug 18. PMID 37934530
- [Derived] Baskerville WA, Friedman TC, Hurley B, Hsieh S, Dixon T, Mtume N, Lee ML, Rodriguez L, Lopez B, Ray LA. Embedding comprehensive smoking cessation programs into community clinics: study protocol for a cluster-randomized controlled trial. Trials. 2022 Feb 3;23(1):109. doi: 10.1186/s13063-022-06023-3. PMID 35115017